CLINICAL TRIAL: NCT04885998
Title: A Phase 1b Study Evaluating the Safety and Efficacy of AMG 757 in Combination With AMG 404 in Subjects With Small Cell Lung Cancer (SCLC)
Brief Title: AMG 757 and AMG 404 in Subjects With Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20200439; 2020-005957-26 (EudraCT Number)
Expanded Access: NCT06064500 (Approved for marketing)
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; SCLC; Lung Cancer; AMG 757; AMG 404; Tarlatamab
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — AMG 757

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose Exploration (Experimental): The recommended phase 2 target dose (RP2D) of tarlatamab in combination with AMG 404 will be estimated using a modified toxicity probability interval (mTPI-2) design. A combination RP2D may be identified based on emerging safety, efficacy, and pharmacodynamic data prior to reaching an maximum tolerated dose (MTD).
  Interventions: Drug: Tarlatamab; Drug: AMG 404
- Phase 2: Dose Expansion (Experimental): Participants will receive the RP2D of tarlatamab in combination with AMG 404 identified in Phase 1 (dose exploration) of the study.
  Interventions: Drug: Tarlatamab; Drug: AMG 404

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab will be administered as an intravenous (IV) infusion.
  Other Names: AMG 757
Drug: AMG 404 — AMG 404 will be administered as an intravenous (IV) infusion.

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, and recommended phase 2 target dose of tarlatamab in combination with AMG 404.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent/assent prior to initiation of any study specific activities/procedures
* Age greater than or equal to 18 years old at the same time of signing the informed consent
* Participants with histologically or cytologically confirmed Small Cell Lung Cancer (SCLC) who progressed or recurred following at least 1 platinum-based regimen
* Eastern Cooperative Oncology Group (ECOG) 0 to 1
* Participants with treated brain metastases are eligible provided they meet defined criteria
* Adequate organ function as defined in protocol

Exclusion Criteria:

* History of other malignancy within the past 2 years with exceptions
* Major surgery within 28 days of first dose of tarlatamab
* Untreated or symptomatic brain metastases and leptomeningeal disease
* Prior anti-cancer therapy, including anti-PD1 or anti-PDL1 antibody therapy: at least 28 days must have elapsed between any prior anti-cancer therapy and the first planned dose of tarlatamab

Exceptions:

* Participants who received prior chemotherapy must have completed at least 14 days before the first dose of tarlatamab and all treatment-related toxicity resolved to grade ≤ 1.
* Participants who received prior palliative radiotherapy must have completed at least 7 days before the first dose of tarlatamab

  * Participants who received prior tarlatamab therapy or prior delta-like ligand 3 (DLL3) x cluster of differentiation 3 (CD3) bispecific therapy are not eligible
  * Participants who experienced recurrent grade 2 pneumonitis or severe or life-threatening immune-mediated adverse events or infusion-related reactions including those that lead to permanent discontinuation while on treatment with immuno-oncology agents
  * History of any immune-related colitis. Infectious colitis is allowed if evidence of adequate treatment and clinical recovery exists and at least 3 months interval observed since diagnosis of colitis
  * Participants with evidence of interstitial lung disease or active, non-infectious pneumonitis
  * Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of tarlatamab
  * History of solid organ transplantation
  * History of hypophysitis or pituitary dysfunction
  * Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study. Participants with Type I diabetes, vitiligo, psoriasis, hypo- or hyper-thyroid disease not requiring immunosuppressive treatment are permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2024-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (7):
  - Northwestern University, Robert H Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Wake Forest Baptist Comprehensive Cancer Research Center, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Austria (2):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- Taiwan (2):
  - Chung Shan Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 research centers in Belgium, Japan, Singapore, Taiwan, and the United States between 27 September 2021 and 11 September 2024. The final analysis data is presented.
Pre-assignment Details: Adults with confirmed diagnosis of small cell lung cancer who progressed or recurred following ≥1 platinum-based treatment regimen were enrolled into sequential dose-exploration (Part 1) and dose-expansion (Part 2) cohorts to receive tarlatamab + AMG 404. Tarlatamab doses ranged from Dose A to Dose D (lowest to highest). The primary outcome measures have been updated, as 1 participant was found post-database lock to have been misclassified in Part 1 (Cohort 3) instead of Part 2.
Groups:
- Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404: Participants received tarlatamab administered intravenously (IV) with 1-step dosing: Dose A on cycle 1 day 1 followed by Dose B on cycle 1 day 8 and cycle 1 day 15, and Dose B Q2W thereafter. Each cycle was 28 days.
  Participants also received a fixed dose short-term infusion of AMG 404 every 28 days.
- Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404: Participants received tarlatamab administered IV with 1-step dosing: Dose A on cycle 1 day 1 followed by Dose C on cycle 1 day 8 and cycle 1 day 15, and Dose C Q2W thereafter. Each cycle was 28 days.
  Participants also received a fixed dose short-term infusion of AMG 404 every 28 days.
- Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404: Participants received tarlatamab administered IV with 1-step dosing: Dose A on cycle 1 day 1 followed by Dose D on cycle 1 day 8 and cycle 1 day 15, and Dose D Q2W thereafter. Each cycle was 28 days.
  Participants also received a fixed dose short-term infusion of AMG 404 every 28 days.
- Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404: Participants received tarlatamab administered IV with 1-step dosing: Dose A on cycle 1 day 1 followed by Dose B on cycle 1 day 8 and cycle 1 day 15, and Dose B Q2W thereafter. Each cycle was 28 days.
  Participants also received a fixed dose short-term infusion of AMG 404 every 28 days.
Period: Overall Study
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404
Started | 7 | 5 | 3 | 8
Safety Analysis Set | 7 | 5 | 3 | 8
Entered Extended Safety Period (EP) | 6 | 1 | 1 | 4
Completed | 3 | 0 | 1 | 3
Not Completed | 4 | 5 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Death | 2 | 1 | 2 | 2
Not completed — Decision by sponsor | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404; Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404: Participants received tarlatamab administered IV with 1-step dosing: Dose A on cycle 1 day 1 followed by Dose B on cycle 1 day 8 and cycle 1 day 15, and Dose B Q2W thereafter. Each cycle was 28 days.
  Participants also received a fixed dose short-term infusion of AMG 404 every 28 days.
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404 | Total
Number analyzed (Participants) | 7 | 5 | 3 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (5.9) | 60.4 (12.7) | 59.3 (18.4) | 55.9 (12.6) | 60.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 5 | 12
  Male | 4 | 2 | 2 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 4 | 1 | 4 | 15
  Unknown or Not Reported | 1 | 1 | 2 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 4 | 1 | 4 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants Who Experienced Dose-limiting Toxicity (DLT)
Description: A DLT was any of the following during the DLT window, assessed by Common Terminology Criteria for Adverse Events v4.0:
  * Grade 3 adverse event (AE) except for fatigue lasting < 7 days, Grade 3 nonfebrile neutropenia that improved to ≤ Grade 1 within 3 weeks, endocrinopathies if managed with replacement therapy, Grade 3 nausea/vomiting or diarrhea for < 72 hours, Grade 3 amylase or lipase values not associated with pancreatitis, Grade 3 hematologic laboratory abnormalities not clinically relevant, or Grade 3 electrolyte abnormality up to 72 hours.
  * Grade 4 AE except for Grade 4 nonfebrile neutropenia lasting ≤ 7 days, Grade 4 electrolyte abnormality lasting up to 72 hours, Grade 4 amylase or lipase values not associated with pancreatitis, or Grade 4 hematologic laboratory abnormalities no clinically relevant.
  * Grade 5 AE
  * Recurrent Grade ≥ 2 pneumonitis
  * Any other toxicity requiring permanent discontinuation of AMG 404.
Time Frame: First dose of tarlatamab up to 28 days
Population: The DLT analysis set included all enrolled participants who received at least 1 dose of tarlatamab or AMG 404 during the dose exploration part of the study with an evaluable DLT endpoint. DLT evaluable endpoints included: 1. participant experienced a DLT; or 2. participant did not experience a DLT and received tarlatamab or AMG 404 treatment as planned in cycle 1 and had been followed for safety events a minimum of 28 days from the date of first dose administration of tarlatamab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404
Number analyzed (Participants) | 6 | 5 | 3
Participants | 0 | 1 | 1

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical trial participant. A TEAE was an AE that started on or after the first dose of investigational product (IP; tarlatamab) up to 65 days after the last dose of tarlatamab or AMG 404 or the end of study (EOS), whichever was earlier. A TEAE for the EP was an AE that occurred after the 65th day after the last dose of tarlatamab or AMG 404 up to 145 days after the last dose of tarlatamab or AMG 404 or end of study, whichever was later. A treatment-related AE was any TEAE where there was a reasonable possibility that the TEAE could have been caused by tarlatamab or AMG 404. Any clinically significant changes in vital signs, physical examinations, electrocardiograms, and clinical laboratory tests were included as TEAEs.
Time Frame: Any TEAEs: From first IP dose up to last dose + 65 days or EOS, median duration was 4.2 months; TEAEs for EP: From last dose + 65 days up to snapshot date (15 November 2024), death, or last dose + 145 days or EOS, median duration was 2.6 months
Population: The safety analysis set included all participants who received at least 1 dose of tarlatamab or AMG 404. For any TEAEs, categories included those that occurred before or during the EP. For the EP, data are presented for participants who entered the EP. Participants with snapshot date (15 November 2024) or death or EOS within the last dose date + 65 days were excluded from the EP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404
Number analyzed (Participants) | 7 | 5 | 3 | 8
Participants
  Any TEAE | 7 | 5 | 3 | 8
  Any tarlatamab-related TEAE | 6 | 5 | 3 | 8
  Any AMG 404-related TEAE | 6 | 4 | 1 | 6
  EP: Any TEAE: number analyzed (Participants) | 6 | 1 | 1 | 4
  EP: Any TEAE | 2 | 0 | 1 | 1
  EP: Any tarlatamab-related TEAE: number analyzed (Participants) | 6 | 1 | 1 | 4
  EP: Any tarlatamab-related TEAE | 1 | 0 | 0 | 0
  EP: Any AMG 404-related TEAE: number analyzed (Participants) | 6 | 1 | 1 | 4
  EP: Any AMG 404-related TEAE | 1 | 0 | 0 | 0

3. Secondary Outcome: Objective Response Rate Per Modified Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: The objective response rate was defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR) based on the modified RECIST v1.1.
  CR: complete disappearance of all lesions and pathologic lymph nodes reduced in short axis to < 10 mm. PR: decrease in tumor burden of ≥ 30% relative to baseline, or complete disappearance of all index lesions with the presence of non-index lesions. Confirmation scans were required within 4 weeks of the first documented response of CR or PR. Exact 95% confidence intervals (CIs) were calculated using the Clopper-Pearson method.
Time Frame: From first dose of IP up to a minimum of last dose date + 65 days or EOS; median (min, max) duration was 4.2 (0.4, 25.4) months
Population: The safety analysis set included all participants who received at least 1 dose of IP (tarlatamab or AMG 404).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404
Number analyzed (Participants) | 7 | 5 | 3 | 8
percentage of participants | 57.1 [18.4 to 90.1] | 20.0 [0.5 to 71.6] | 66.7 [9.4 to 99.2] | 37.5 [8.5 to 75.5]

4. Secondary Outcome: Duration of Response Per Modified RECIST v1.1
Description: The duration of response was defined as the time from first evidence of CR or PR to progressive disease (PD) or death due to any cause, whichever occurred first, estimated via Kaplan-Meier methods.
  CR: complete disappearance of all lesions and pathologic lymph nodes reduced in short axis to < 10 mm. PR: decrease in tumor burden of ≥ 30% relative to baseline, or complete disappearance of all index lesions with the presence of non-index lesions. Confirmation scans were required within 4 weeks of the first documented response of CR or PR. PD: radiologic detection of ≥ 20% increase in tumor burden relative to nadir and ≥ 5 mm absolute increase, or unequivocal progression of non-index lesions, or presence of new lesions. 95% CIs were calculated using the Brookmeyer and Crowley method.
Time Frame: as for outcome 3
Population: The safety analysis set included all participants who received at least 1 dose of IP (tarlatamab or AMG 404). Data is presented for participants who achieved a best overall response of PR or CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404
Number analyzed (Participants) | 4 | 1 | 2 | 3
months | NA [3.9 to NA] — Median and upper confidence interval (CI) were not calculable as median was not reached due to insufficient event data occurring. | 6.0 [NA to NA] — Upper and lower CIs were not calculable due to only 1 participant achieving OR. | 8.1 [4.7 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | 11.2 [5.6 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median.

5. Secondary Outcome: Disease Control Rate Per Modified RECIST v1.1
Description: The disease control rate was defined as the percentage of participants with a best overall response of a confirmed response (CR/PR) or stable disease (SD) while on the study as defined by modified RECIST v1.1.
  CR: complete disappearance of all lesions and pathologic lymph nodes reduced in short axis to < 10 mm. PR: decrease in tumor burden of ≥ 30% relative to baseline, or complete disappearance of all index lesions with the presence of non-index lesions. Confirmation scans were required within 4 weeks of the first documented response of CR or PR SD: Index lesions not meeting the criteria for CR, PR, or PD or the persistence of one or more non-index lesions. Exact 95% CIs were calculated using the Clopper-Pearson method.
Time Frame: as for outcome 3
Population: The safety analysis set included all participants who received at least 1 dose of IP (tarlatamab or AMG 404).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404
Number analyzed (Participants) | 7 | 5 | 3 | 8
percentage of participants | 57.1 [18.4 to 90.1] | 60.0 [14.7 to 94.7] | 66.7 [9.4 to 99.2] | 50.0 [15.7 to 84.3]

6. Secondary Outcome: Progression-free Survival Per Modified RECIST v1.1
Description: Progression-free survival was defined as the interval from the earlier date of the first dose of IP to the earlier of PD per modified RECIST v1.1 or death due to any cause, estimated via Kaplan-Meier methods.
  PD: radiologic detection of ≥ 20% increase in tumor burden to nadir and ≥ 5 mm absolute increase, or unequivocal progression of non-index lesions, or the presence of new lesions.
  Confirmation scans were required within 4 weeks of the first documented response of CR or PR, and 4-6 weeks for PD. 95% CIs were calculated using the Brookmeyer and Crowley method.
Time Frame: From first dose of IP up to a minimum of EOS or death; median (min, max) time was 9.4 (0.4, 25.5) months
Population: The safety analysis set included all participants who received at least 1 dose of IP (tarlatamab or AMG 404).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404
Number analyzed (Participants) | 7 | 5 | 3 | 8
months | 6.5 [0.4 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | 3.8 [1.8 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | 6.5 [3.0 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | 7.4 [1.6 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median.

7. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval from the earlier date of the first dose of IP to the event of death due to any cause, estimated via Kaplan-Meier methods. Participants who were still alive were censored at the date last known to be alive. If the date last known to be alive was after the data cutoff date, the participant was censored at the analysis trigger date. 95% CIs were calculated using the Brookmeyer and Crowley method.
Time Frame: From first dose of IP up to a minimum of EOS or death; median (min, max) time was 9.4 (0.4, 25.5) months
Population: The safety analysis set included all participants who received at least 1 dose of IP (tarlatamab or AMG 404).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404
Number analyzed (Participants) | 7 | 5 | 3 | 8
months | NA [0.4 to NA] — Median and upper confidence interval (CI) were not calculable as median was not reached due to insufficient event data occurring. | NA [2.7 to NA] — Median and upper confidence interval (CI) were not calculable as median was not reached due to insufficient event data occurring. | 6.5 [3.0 to NA] — Upper CI was not calculable due to insufficient event data occurring above the median. | NA [4.8 to NA] — Median and upper confidence interval (CI) were not calculable as median was not reached due to insufficient event data occurring.

8. Secondary Outcome: Maximum Observed Concentration (Cmax) of Tarlatamab in Combination With AMG 404
Description: Cmax was obtained using noncompartmental analysis, which was performed for tarlatamab PK parameter estimation. PK analysis is presented per dose received as pre-specified.
Time Frame: Cycle 2 Day 1 (pre-dose up to 7 days post-dose); Cycle 2 Day 15 (pre-dose up to 14 days post-dose)
Population: The pharmacokinetic (PK) analysis set included all participant who had received at least 1 dose of tarlatamab and had at least 1 PK sample collected. Participants with data available at each timepoint are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Groups:
- PK Analysis: Tarlatamab Dose B + AMG 404: Participants received tarlatamab administered IV with Dose B on cycle 1 day 8 and cycle 1 day 15, and Dose B Q2W thereafter. Each cycle was 28 days.
  Participants also received a fixed dose short-term infusion of AMG 404 every 28 days.
- PK Analysis: Tarlatamab Dose C + AMG 404: Participants received tarlatamab administered IV with Dose C on cycle 1 day 8 and cycle 1 day 15, and Dose C Q2W thereafter. Each cycle was 28 days.
  Participants also received a fixed dose short-term infusion of AMG 404 every 28 days.
- PK Analysis: Tarlatamab Dose D + AMG 404: Participants received tarlatamab administered IV with Dose D on cycle 1 day 8 and cycle 1 day 15, and Dose D Q2W thereafter. Each cycle was 28 days.
  Participants also received a fixed dose short-term infusion of AMG 404 every 28 days.
Arm/Group | PK Analysis: Tarlatamab Dose B + AMG 404 | PK Analysis: Tarlatamab Dose C + AMG 404 | PK Analysis: Tarlatamab Dose D + AMG 404
Number analyzed (Participants) | 12 | 4 | 1
micrograms per milliliter
  Cycle 2 Day 1 | 2.98 (37) | 8.12 (28) | 28.1 (NA) — Geometric coefficient of variation was not calculable due to only 1 participant having available data
  Cycle 2 Day 15: number analyzed (Participants) | 10 | 4 | 1
  Cycle 2 Day 15 | 3.29 (40) | 5.54 (64) | 21.2 (NA) — Geometric coefficient of variation was not calculable due to only 1 participant having available data

9. Secondary Outcome: Trough Concentration (Ctrough) of Tarlatamab in Combination With AMG 404
Description: Ctrough was obtained at the end of a dosing interval or just before the administration of the next planned dose using noncompartmental analysis, which was performed for tarlatamab PK parameter estimation. PK analysis is presented per dose received as pre-specified.
Time Frame: Cycle 2 Day 15 (pre-dose)
Population: PK analysis set included all participant who had received at least 1 dose of tarlatamab and had at least 1 PK sample collected. Participants with data available are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | PK Analysis: Tarlatamab Dose B + AMG 404 | PK Analysis: Tarlatamab Dose C + AMG 404 | PK Analysis: Tarlatamab Dose D + AMG 404
Number analyzed (Participants) | 6 | 4 | 1
micrograms per milliliter | 0.380 (27) | 0.893 (37) | 6.59 (NA) — Geometric coefficient of variation was not calculable due to only 1 participant having available data

10. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 336 Hours (AUC0-336) of Tarlatamab in Combination With AMG 404
Description: AUC0-336 was defined as the actual body exposure to the drug over time following administration of a dose, calculated from time zero to 336 hours post-dose using noncompartmental analysis, which was performed for tarlatamab PK parameter estimation. PK analysis is presented per dose received as pre-specified.
Time Frame: Cycle 2 Day 1 (pre-dose up to 7 days post-dose); Cycle 2 Day 15 (pre-dose up to 14 days post-dose)
Population: PK analysis set included all participant who had received at least 1 dose of tarlatamab and had at least 1 PK sample collected. Participants with data available at each timepoint are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*micrograms per milliliter
Arm/Group | PK Analysis: Tarlatamab Dose B + AMG 404 | PK Analysis: Tarlatamab Dose C + AMG 404 | PK Analysis: Tarlatamab Dose D + AMG 404
Number analyzed (Participants) | 11 | 4 | 1
hours*micrograms per milliliter
  Cycle 2 Day 1 | 378 (39) | 1060 (31) | 4180 (NA) — Geometric coefficient of variation was not calculable due to only 1 participant having available data
  Cycle 2 Day 15: number analyzed (Participants) | 9 | 4 | 1
  Cycle 2 Day 15 | 336 (37) | 621 (72) | 3950 (NA) — Geometric coefficient of variation was not calculable due to only 1 participant having available data

ADVERSE EVENTS:
Time Frame: For all-cause mortality, from enrollment to study completion; median time on study was 9.4 (0.4, 25.5) months. TEAEs were collected from first dose of IP up to last dose + 65 days or EOS; median (min, max) duration was 4.2 (0.4, 25.4) months. TEAEs for the EP were collected from 65 days up to 145 days or EOS after the last dose of tarlatamab or AMG 404; median (min, max) duration was 2.6 (0.6, 8.4) months.
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all participants enrolled in the study.
  Participants with snapshot date (15 November 2024) or death or EOS within the last dose date + 65 days were excluded from the EP.
Groups:
- Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 (EP): Participants in Part 1 Cohort 1 who entered the EP from 65 days up to 145 days or EOS after the last dose of tarlatamab or AMG 404.
- Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 (EP): Participants in Part 1 Cohort 2 who entered the EP from 65 days up to 145 days or EOS after the last dose of tarlatamab or AMG 404.
- Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 (EP): Participants in Part 1 Cohort 3 who entered the EP from 65 days up to 145 days or EOS after the last dose of tarlatamab or AMG 404.
- Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404 (EP): Participants in the Part 2 Dose Expansion Cohort who entered the EP from 65 days up to 145 days or EOS after the last dose of tarlatamab or AMG 404.
- Part 2 Dose Expansion Cohort: Tarlatamab Dose A/B + AMG 404: Participants received tarlatamab administered IV with 1-step dosing: Dose A on cycle 1 day 1 followed by Dose B on cycle 1 day 8 and cycle 1 day 15, and Dose B Q2W thereafter. Each cycle was 28 days. Participants also received a fixed dose short-term infusion of AMG 404 every 28 days.
Arm/Group | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 (EP) | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 (EP) | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 (EP) | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404 (EP) | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/B + AMG 404
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/6 | 1/5 | 0/1 | 1/3 | 1/1 | 2/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 5/7 | 1/6 | 3/5 | 0/1 | 2/3 | 1/1 | 0/4 | 5/8
Other Adverse Events (participants affected / at risk) | 7/7 | 1/6 | 5/5 | 0/1 | 2/3 | 0/1 | 1/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 (N=7) | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 (EP) (N=6) | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 (N=5) | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 (EP) (N=1) | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 (N=3) | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 (EP) (N=1) | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404 (EP) (N=4) | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/B + AMG 404 (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 (N=7) | Part 1 Cohort 1: Tarlatamab Dose A/Dose B + AMG 404 (EP) (N=6) | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 (N=5) | Part 1 Cohort 2: Tarlatamab Dose A/Dose C + AMG 404 (EP) (N=1) | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 (N=3) | Part 1 Cohort 3: Tarlatamab Dose A/Dose D + AMG 404 (EP) (N=1) | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/Dose B + AMG 404 (EP) (N=4) | Part 2 Dose Expansion Cohort: Tarlatamab Dose A/B + AMG 404 (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 3
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 3 | 0 | 2 | 0 | 1 | 0 | 0 | 2
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 5
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight loss poor (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urinary tract discomfort (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood prolactin abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT04885998/Prot_002.pdf
  • Statistical Analysis Plan (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT04885998/SAP_003.pdf